CLINICAL TRIAL: NCT06432764
Title: A Phase Ib Open Label Positron Emission Tomography Study to Assess Changes in Intestinal [11C]AZ14132516 Uptake Following Administration of Multiple Doses of AZD7798 to Patients With Crohn's Disease.
Brief Title: Positron Emission Tomography Study of Changes in [11C]AZ14132516 Uptake Following Administration of AZD7798 to Patients With Crohn's Disease.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9690C00007; 2024-512992-11-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Drug Evaluation; Radioligand Assay

STUDY DESIGN:
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD7798 (Experimental): Arm consists of up to 2 panels
  Interventions: Drug: AZD7798; Drug: [11C]AZ14132516

INTERVENTIONS:
Drug: AZD7798 — Each participating patient will receive the study drug as specified in the study protocol.
  Other Names: Study Drug
Drug: [11C]AZ14132516 — A single microdose (≤ 10 μg) of radiopharmaceutical [11C]AZ14132516 will be extemporaneously prepared and administered to each participant prior to each PET examination
  Other Names: Radioligand

SUMMARY:
The purpose of this study is to measure the changes in intestinal uptake of radioligand [11C]AZ14132516 following multiple doses of AZD7798 in participants with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 20 to 80 years of age, inclusive, at the time of signing the informed consent.
* Participants with confirmed Crohn's disease with small bowel involvement (Montreal terminal ileum [L1] or ileocolon [L3]) per study gastroenterologist (diagnosed via combination of clinical findings and at least one of endoscopy and/or histology and/or imaging) with diagnosis made at least 6 months before screening.
* Participants with active Crohn's disease as determined by one of the following:

  1. Evidence of active inflammation on cross-sectional imaging (CT, MRI or bowel ultrasound scan) or endoscopy within 6 months before screening OR EITHER
  2. If no cross-sectional imaging or endoscopy performed within 6 months before screening, a bowel ultrasound scan may be performed to confirm active disease OR
  3. If no cross-sectional imaging or endoscopy performed within 6 months before screening, elevated faecal calprotectin AND CRP
* Body habitus compatible with PET examination.
* Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent
* Able and willing to participate in all scheduled evaluations, abide by all study restrictions, and complete all required tests and procedures.

Exclusion Criteria:

* Other form of IBD or concomitant, additional, active GI luminal inflammatory diseases.
* CMV colitis within 12 months before screening.
* Crohn's complications including short bowel syndrome, strictures that are symptomatic or with pre-stenotic dilatation or other conditions where surgery anticipated during study period.
* Planned bowel or perianal surgery within 6 months before screening.
* Bowel resection surgery within 6 months before screening.
* Undrained fistula or abscess (including active perianal disease).
* Positive Clostridium difficile toxin test during screening.
* Current significant major or unstable respiratory disease, heart disease, cerebrovascular disease, haematological disease, hepatic disease, renal disease, GI disease, or other major diseases other than active Crohn's disease and associated extra-intestinal manifestations.
* Ongoing psychiatric conditions that in the opinion of the Investigator, precludes study participation.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to biologic therapies.
* Participants with unstable hypertension (as judged by the Investigator) or symptomatic hypotension, history of pre-syncope or syncope due to orthostatic hypotension and/or induced by change of posture.
* Significant abnormalities on clinical examination, including neurological and physical examination, vital signs, and ECG, other than signs of Crohn's disease.
* Clinical chemistry, haematology, or urine analysis results that may interfere with the study or present a safety risk to the participant.
* Abnormal vital signs, after 10 minutes of supine rest as judged by the Investigator.
* Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG that may interfere with the interpretation of QTc changes.
* Positive hepatitis B, hepatitis C, or HIV serology
* Treatment with an anti-TNF within 8 weeks of the first dose and throughout the study period, before the first dose and throughout study period, unless therapeutic drug monitoring is performed, and drug concentrations are undetectable.
* Treatment with any biologic, other than an anti-TNF (including vedolizumab and ustekinumab) within 12 weeks prior to first dose and throughout the study period, unless therapeutic drug monitoring is performed, and drug concentrations are undetectable.
* Treatment with rituximab within 12 months before first dose and throughout the study period.
* Treatment with Sphigosine-1-phosphate receptor modulators or Janus kinase inhibitors within 4 weeks before first dose and throughout the study period.
* Treatment with apheresis (eg, Adacolumn, Cellsorba) within 2 weeks prior to first dose and throughout the study period.
* Treatment with corticosteroids at a total daily dose of greater than 20 mg prednisone or equivalent (greater than 9 mg budesonide).
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or site staff).
* Judgement by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
* Suffers from claustrophobia that limits the ability to undergo the scanning procedure.
* Positive SARS-CoV-2 rapid antigen test at screening.
* Any other reason that, in the study Investigator opinion, prohibits the inclusion of the participants into the study.
* Judgement by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
* Live or attenuated vaccine within 4 weeks before screening and until 12 weeks after the end of the follow-up period (1 year for Bacillus Calmette-Guérin vaccination).
* An active infection, or history of serious infection within 28 days before screening.
* History of symptomatic herpes simplex (excluding cold sores) or herpes zoster infection within 3 months prior to screening.
* Positive or indeterminate TB QuantiFERON test performed within 1 year of screening (without known interval exposure to TB) or during screening period unless evidence of completion of full treatment course for latent TB with no clinical symptoms or signs indicative of re activation.
* Chest x-ray with signs of malignancy or latent or active TB infection performed within 1 year of screening (without known interval exposure to TB) or during screening period.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days/5 half-lives, whichever is longer, of the first administration of IMP in this study. The period of exclusion begins 30 days/5 half-lives after the final dose, whichever is longer, .
* Current malignancy or history of malignancy, except for:

  1. Basal cell carcinoma, localised squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the participant is in remission and curative therapy was completed at least 12 months prior to screening.
  2. Other non-GI malignancies are eligible provided that the participant is in remission and curative therapy was completed at least 5 years before screening.
* For females only: Currently pregnant (confirmed with positive pregnancy test) or breastfeeding.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-04-16 (Estimated); Study Completion 2026-04-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in intestinal SUV/SUVR | Weeks 13, 16, 20 and 24 (may vary between participants)
  Standardized uptake value (SUV) is the radioactivity concentration in given region of interest normalized for injected radioactivity and body weight.
  Standardised uptake value ratio (SUVR) is the ratio of SUV in a given region of interest to a reference region without significant radioligand uptake

SECONDARY OUTCOMES:
Serum AZD7798 concentration | Weeks 0, 4, 8, 12 (may vary between participants)
Incidence and titre of anti-drug antibodies | Week 0, 4, 8, 12 and 24 (may vary between participants)

OTHER OUTCOMES:
Number of participants with safety findings, AEs | Until final follow-up, week 24 (may vary between participants)
  Safety will be assessed by Adverse Events, vital signs, haematology and clinical chemistry

CONTACTS AND LOCATIONS:
Overall Officials: Maria Creignou, Principal Investigator — Karolinska University Hospital
Locations (1):
- Research Site, Stockholm, Sweden